CLINICAL TRIAL: NCT06954558
Title: The Phase I, Open-label, Single-arm Clinical Study Evaluating the Safety, Pharmacokinetics, and Preliminary Efficacy of GK01 Cell Injection in Patients With Advanced Solid Tumors
Brief Title: A Single-Arm, Open-Label, Phase I Study of GK01 for Advanced Solid Tumor
Acronym: GUARDIAN
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Collaborators: Beijing Geek Gene Technology Co., LTD (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GK01IIT-TZ01
Record Dates: First submitted 2025-04-14; First posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-03

CONDITIONS: Advanced Solid Tumors
Keywords: efficacy; safety; PK; TILs

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GK01 injection (Experimental): Autologous tumor-reactive T cells injection
  Interventions: Drug: GK01 Injection

INTERVENTIONS:
Drug: GK01 Injection — Autologous tumor-reactive T cells injection

SUMMARY:
This study is a Phase I, open-label, single-arm clinical trial to evaluate the safety, pharmacokinetics, and preliminary efficacy of GK01 in patients with advanced solid tumors.

ELIGIBILITY:
1. Ability to understand and sign a written informed consent document；
2. At the date of signing ICF, 18 ~70 years old, male or female；
3. Histopathological confirmed advanced solid tumor patients who have failed to standard treatment or intolerance with standard treatment；
4. There is at least one resectable tumor lesion that has not received radiation therapy or other local therapies;
5. At least one measurable lesion at baseline per RECIST version 1.1；
6. The expected survival time is more than 12 weeks;
7. ECOG 0-1 points;
8. Adequate organ functions

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-03-18 (Actual); Primary Completion 2028-03-18 (Estimated); Study Completion 2028-07-18 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | 2 years
  The incidence and severity, and correlation of AEs (Adverse Events) and SAEs (Serious Adverse Events).

SECONDARY OUTCOMES:
PK | 2 years
  Levels of T-cell Receptor copies
Objective response rate (ORR) | 2 years
Progress-free survival(PFS) | 2 years
  PFS will be assessed from the first GK01 infusion to death from any cause or the first assessment of progression (Assessed based on RECIST criteria)
Overall survival (OS ) | 2 years
  OS will be assessed from the first GK01 infusion to death from any cause (Assessed based on RECIST criteria)
Disease control rate (DCR) | 2 years
Patient Quality of Life | 2 years
  EORTC(European Organisation for Research and Treatment of Cancer) QLG (Quality of Life Group)Core Questionnaire (EORTC QLQ-C30)
PD marker | 2 years
  Concentration levels of serum cytokines, such as IL-2, IL-4, IL-6, IL-10, IFN-γ, TNF-α

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute & Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No